CLINICAL TRIAL: NCT00542711
Title: Liquid Tumeric Extract for Increasing Bio-availability of Curcumin in the Human Body: Pharmacokinetic Study.
Brief Title: Bio-availability of a New Liquid Tumeric Extract
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Technical difficulties
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Hadassah Medical Organization, Hadassah Medical Organization
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Curcumol-HMO-CTIL
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Curcumin; Bioavilability; Healthy subjects
MeSH Terms: interventions — Curcumin; curcumol

INTERVENTIONS:
Drug: liquid tumeric/curcumin extract — 30 drops (4 participants), 50 drops (4 participants) and 70 drops (4 participants). one dose.
  Other Names: Curcumol (patent pending, Israel Patent Application No. 181,121).

SUMMARY:
Curcumin is a commonly-used spice and food coloring. Evidence suggests that curcumin can suppress tumor initiation, promotion and metastasis in a variety of tumor cell lines. The current available curcumin has low bioavailability restricting the effect of curcumin in non-colon cancer. In this study we plan to test a new liquid tumeric/curcumin extract, Curcumol (patent pending, Israel Patent Application No. 181,121). We predict the bioavailability of the liquid tumeric/curcumin extract will be better compared to the currently used curcumin powder.

DETAILED DESCRIPTION:
Twelve healthy participants enrolled to the study. All volunteers will have pre study evaluation to confirm healthy state. After enrollment, each participant will be tested twice, one with the liquid tumeric/curcumin (study drug) and once with the curcumin powder (control). The days of testing will be on two days, separated by two weeks wash-out period. The participants will be assigned to randomly receive study drug or control on the 1st day, with the other regimen administered at the 2nd day. Both study drug and control will be diluted in 150ml of water. The doe of study drug will be escalated from 30 drops (4 participants), 50 drops (4 participants) and 70 drops (4 participants). Blood sample will be collected at 0,0.25,0.5,0.75,1,2,3,4,5,6,8h post drug. Quantization of curcumin plasma levels will be done by the high pressure liquid chormatography method. A biomarker for the potential effect of curcumin, platelet function pre and post curcumin consumption will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Complete Healthy
* Able to attend two full days of study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shoshana Revel-Vilk, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel